CLINICAL TRIAL: NCT02413502
Title: Collection and Storage of Biological Samples Obtained by Leukapheresis for the Future Study of Immune Responses After BCG Vaccination in BCG-naïve Healthy Adults in the US (A-046)
Brief Title: Leukapheresis Sampling for Immune Responses After BCG Vaccination in BCG-naïve Healthy Adults in the US
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Aeras (Other)
Collaborators: University of Rochester (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: A-046
Record Dates: First submitted 2015-03-10; First posted 2015-04-10 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2015-10

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis | interventions — BCG Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bacillus Calmette-Guérin (BCG) (Experimental): Tice brand BCG used to vaccinate BCG-Naïve adults.
  Interventions: Biological: BCG

INTERVENTIONS:
Biological: BCG — BCG Vaccine USP attenuated live culture for percutaneous use (Merck) at 1-8 x 10^8 CFUs.
  Other Names: TICE BCG

SUMMARY:
The objective of this protocol is to obtain biological samples through leukapheresis and cryopreservation of cells for the future study, by in vitro assay, of immune responses after one dose of BCG in BCG-naïve healthy adults.

DETAILED DESCRIPTION:
This is an open-label protocol in 12 healthy adults who are BCG-naïve. All participants will receive a single dose of BCG, by percutaneous administration, on Study Day 0. There will be two follow-up visits on Study Days 54 and 56, with telephone contact every 2 weeks in between these visits. Leukapheresis will be conducted on Study Days 0 and 56. The Study Day 56 leukapheresis was selected based on results from functional biological assays that suggest analysis of samples at this time point may provide insight into the protective immune responses elicited by BCG. The study will be conducted at a single site in the US (University of Rochester Medical Center [URMC]).

ELIGIBILITY:
Inclusion Criteria:

1. Has completed the written informed consent process.
2. Is age ≥18 years and ≤55 years on Study Day 0.
3. Agrees to stay in contact with the study site for the duration of the study, provide updated contact information as necessary, and has no current plans to move from the study area for the duration of the study.
4. Agrees to avoid elective surgery during the study.
5. Willingness to receive HIV test results.
6. For female participants: agrees to avoid pregnancy from 21 days prior to Study Day 0 and for the full duration of the study.
7. Has general good health, confirmed by medical history and physical examination.
8. Has not received vaccination or immunotherapy with a BCG product at any time prior to Study Day 0.

Exclusion Criteria:

1. Acute illness on Study Day 0.
2. HIV-1/2 positive
3. Oral temperature ≥37.5°C on Study Day 0.
4. Abnormal laboratory values per local laboratory parameters from most recent blood collection prior to Study Day 0 for specific parameters listed in the protocol.
5. Evidence of significant active infection.
6. Evidence of central nervous system tuberculosis or pleural tuberculosis.
7. Screening TST reaction >5 mm.
8. History of treatment for active or latent tuberculosis infection.
9. History or evidence of active tuberculosis.
10. Shared a residence within the last year with an individual on anti-tuberculosis treatment or with culture or smear positive tuberculosis.
11. History of occupational exposure to an individual with active tuberculosis in a health care setting.
12. History of autoimmune disease or immunosuppression.
13. Used immunosuppressive medication within 42 days before Study Day 0 (inhaled and topical corticosteroids are permitted).
14. Received immunoglobulin or blood products within 42 days before Study Day 0.
15. Received any investigational drug or investigational vaccine within 182 days before Study Day 0, or planned participation in any other interventional study during the study period.
16. Received investigational TB vaccine at any time.
17. Planned administration/administration of a licensed vaccine in the period starting 28 days before and ending 56 days after BCG vaccination in this study.
18. Current chronic drug therapy including hormone replacement such as thyroxin, insulin, etc (estrogen and progesterone replacement and contraceptives are acceptable).
19. History or laboratory evidence of any past, present, or future possible immunodeficiency state including but not limited to any laboratory indication of HIV-1 infection.
20. No contraindications for BCG administration as described in the BCG package insert (Appendix B).
21. Previous medical history that may compromise the safety of the participant in the study, including but not limited to: severe impairment of pulmonary function from tuberculosis infection or other pulmonary disease; chronic illness with signs of cardiac or renal failure; suspected progressive neurological disease; or uncontrolled epilepsy.
22. Evidence of a new acute illness that may compromise the safety of the participant in the study.
23. History or evidence of chronic hepatitis.
24. History of alcohol or drug abuse within the past 2 years.
25. History of keloid formation.
26. Positive urine test for illicit drugs (opiates, cocaine, amphetamines).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2015-05; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Immune response measured by Intracellular cytokine staining (ICS) | Day 56 of the study
  ICS used to characterize the response to BCG.

CONTACTS AND LOCATIONS:
Overall Officials: Ann M. Ginsberg, MD, PhD, Study Director — Aeras